CLINICAL TRIAL: NCT01574612
Title: An Open Label Multi Center Phase III Subject/Caregiver Initiated Safety Study of Xerese(Acyclovir and Hydrocortisone)Cream 5%/1% in the Treatment of Recurrent Herpes Labialis in Children
Brief Title: Open Label Safety Study of Xerese Cream in the Treatment of Recurrent Herpes Labialis in Children 6-11 Years Old
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Meda Pharmaceuticals (Industry)
Collaborators: TKL Research, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP 800
Record Dates: First submitted 2012-04-05; First posted 2012-04-10 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Herpes Labialis
Keywords: Xerese; acyclovir hydrocortisone cream; herpes labialis; pediatric
MeSH Terms: conditions — Herpes Labialis | interventions — Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- topical cream acyclovir/hydrocortisone (Experimental): topical cream acyclovir/hydrocortisone used
  Interventions: Drug: acyclovir/hydrocortisone cream

INTERVENTIONS:
Drug: acyclovir/hydrocortisone cream — cream applied topically to lesion five times daily for five days
  Other Names: Xerese(r)

SUMMARY:
To test the safety of Xerese (acyclovir and hydrocortisone)Cream 5%/1% for the treatment of recurrent cold sores in children ages 6-11yrs after 5 days of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, age 6-11 years at time of enrollment
* General good health, as judged by the Investigator
* History of recurrent herpes labialis with at least two (2) recurrences during the last twelve (12) months, as based on interview with the subject or subject's caregiver
* Agreement to refrain from using other topical medical, over-the counter (OTC), or cosmetic products in or around the oral area during the herpes recurrence
* Agreement to refrain from mechanical disruption of the area affected by herpes labialis during the study recurrence
* Subjects and their legally acceptable representative(s) must voluntarily sign and date the informed assent (subject) and consent (legally authorized representative).
* Willingness to comply with all requirements of the study.

Exclusion Criteria:

* Any evidence of an immunosuppressed state of the subject due to underlying disease (e.g. HIV infection) or concomitant treatment (e.g. cancer chemotherapy)
* Significant skin conditions that occur in the area typically affected by herpes recurrences, and that would interfere with assessment of lesions such as atopic dermatitis, acne, eczema, psoriasis or chronic vesiculobullous disorders
* Administration of an investigational drug or within 30 days prior to inclusion, or concurrent participation in another research study
* Administration of an immunomodulatory agent within the past 30 days
* History of immediate hypersensitivity or serum sickness reaction to any nucleoside analog antiviral agent, or to any topical steroid, or to the vehicle
* Clinically relevant abnormal physical findings at screening which, in the opinion of the investigator, would interfere with the objectives of the study or that may preclude compliance with the study procedures Nursing or pregnant (Pubescent females require pregnancy testing)

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 54 (Actual)
Dates: Start 2012-03; Primary Completion 2012-12 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Ginsburg, D.O., Study Director — Meda Pharma US
Locations (10):
- United States (10):
  - MCS Clinical Trials, Los Angeles, California
  - Sunshine Research Center, Opa-locka, Florida
  - Altus Rsearch,INC, West Palm Beach, Florida
  - Provident Clincal Research, Addison, Illinois
  - Central Kentucky Research, Lexington, Kentucky
  - Rochester Clinical Research, Rochester, New York
  - PGM Research of Winston-Salem, LLC, Winston-Salem, North Carolina
  - Clinical Partners LLC, Johnston, Rhode Island
  - Corsicana Medical Research,PNC, Corsicana, Texas
  - National Clinical Research-Richmond,Inc., Richmond, Virginia

RESULTS

PARTICIPANT FLOW:
Groups:
- Topical Cream: commercial product being used
  acyclovir/hydrocortisone cream: cream applied topically to lesion five times daily for five days
Period: Overall Study
Arm/Group | Topical Cream
Started | 54 (patients who were identified as having the appropriate medical history of herpes labialis)
Completed | 46
Not Completed | 8
Not completed — Adverse Event | 3
Not completed — non compliant with drug | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 2

BASELINE CHARACTERISTICS:
Groups:
- Topical Cream: xerese topical cream is the only active used in this trial
Arm/Group | Topical Cream
Number analyzed (Participants) | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.1 (1.7)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 54
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 31
  Male | 23
Region of Enrollment [Number; unit: participants]
  United States | 54
age of subjects with prior history of herpes labialis outbreak [Number; unit: participants]
  less than or equal to 3 years | 27 (33)
  age 4 to 6 years | 17 (21.5)
  age 7 to 9 years | 10 (13.9)

OUTCOME MEASURES:

1. Primary Outcome: Reporting of Adverse Events
Description: treatment period is for 5 days and follow up visits at 7days and 21 days after first dose
Time Frame: day 1 to day 21
Measure: Number; unit: participants
Groups:
- Topical Cream: commercial cream used
Arm/Group | Topical Cream
Number analyzed (Participants) | 54
participants | 9

ADVERSE EVENTS:
Arm/Group | Topical Cream
Serious Adverse Events (participants affected / at risk) | 0/54
Other Adverse Events (participants affected / at risk) | 9/54
OTHER ADVERSE EVENTS (reported when occurring in more than 1.9% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Topical Cream (N=54)
general disorder (General disorders) | 1
URI (Infections and infestations) | 3
lip injury (Injury, poisoning and procedural complications) | 2
paresthesia oral (Gastrointestinal disorders) | 1
rash (Skin and subcutaneous tissue disorders) | 1
headache (Nervous system disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No